CLINICAL TRIAL: NCT02954016
Title: Safety and Efficacy of the ValenTx EndoPass™ System for the Treatment of Obese Subjects: The ePass Clinical Trial
Brief Title: The ePass Clinical Trial for the Treatment of Obese Subjects
Acronym: ePass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ValenTx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP 1.0
Record Dates: First submitted 2016-09-23; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss; Hypertension; Type 2 Diabetes Mellitus; Hyperlipidemia
MeSH Terms: conditions — Obesity; Weight Loss; Hypertension; Diabetes Mellitus, Type 2; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ePass (Experimental): Subjects implanted with the investigational ValenTx Endo Bypass System
  Interventions: Device: ePass

INTERVENTIONS:
Device: ePass — Subject is implanted with the device for up to 3 years.
  Other Names: ValenTx; Endo Bypass System; EBS

SUMMARY:
To evaluate the safety and efficacy of the endoscopically implanted ValenTx EndoPass™ System for treatment of adults with severe obesity.

The EndoPass System is indicated for weight loss in adults with a body mass index (BMI) ≥35 and ≤ 50 kg/m2 who have failed more conservative weight loss methods.

DETAILED DESCRIPTION:
* Single-arm, multi-center study conducted in up to 50 subjects at up to 5 sites.
* Subjects will be implanted with the EndoPass device for up to 36 months.
* Body weight, adverse events and device function will be monitored at monthly visits for the first year after implant and quarterly visits thereafter.
* Additional follow-up data will include vital signs, hip and waist circumference, blood lab tests, endoscopic and esophagram assessments of the condition of the implanted device, quality of life and eating behavior questionnaires.
* All subjects will be followed for 12 months after device removal.
* A single device renewal may take place as needed after the initial implant.
* Subject study participation may last up to four years, but is expected to vary with implant duration, which will be determined on a case-by-case basis.

ELIGIBILITY:
Key Inclusion Criteria:

* 18-60 years of age.
* BMI ≥ 35 and ≤ 50 kg/m2
* Documented failure with non-surgical weight loss methods
* Self-reported maximum and minimum body weights during the past 12 months within 10% of current body weight

Key Exclusion Criteria:

* Pregnancy or intention of becoming pregnant.
* Past history of esophageal, gastric or bariatric surgery.
* Medical conditions contraindicating elective endoscopic or bariatric procedures.
* Insulin-dependent diabetes mellitus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2021-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects affected by serious adverse device effects (SADEs) as defined by International Standards Organization (ISO) standard 14155:2011. | 1 Year
  The proportion of subjects affected by SADEs during the 12 months following their device implant

SECONDARY OUTCOMES:
12 Month Weight Loss in Kilograms | 1 Year
  Mean reduction in bodyweight in kilograms from the day of implant to the 12 month post-implant follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Maude-Griffin, Study Director — ValenTx, Inc.
Locations (2):
- Hospital Italiano de Mendoza / Clinica Quiriurgica, Mendoza, Argentina
- Swiss Hospital / Especialidades Bariatrices, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No